CLINICAL TRIAL: NCT06196190
Title: The Prognostic Value of Conization and Negative HPV Typing After Conization Prior to Surgical Intervention in Adenocarcinoma in Situ and Early Stage Cervical Cancer
Brief Title: Prognostic Value of Conization and Negative HPV After Conization in AIS and Early Stage Cervical Cancer
Status: Recruiting | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Yoav Siegler B.Sc. M.D, Resident at the Gynecological Oncology Department, Rambam Health Care Campus
Other Study IDs: 0256-23-RMB
Record Dates: First submitted 2023-09-30; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Cervix Cancer; HPV-Related Malignancy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cervical swap for presence of Human papillomavirus DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Post Conization HR HPV positive: Women with a Post Conization cervical test positive for HR HPV
- Post Conization HR HPV negative: Women with a Post Conization cervical test negative for HR HPV
- No Conization HR HPV positive: Women who did not go through Conization prior to surgery and had a cervical test positive for HR HPV
- No Conization HR HPV negative: Women who did not go through Conization prior to surgery and had a cervical test negative for HR HPV

SUMMARY:
In women with cervical cancer -Squamous cell carcinoma, Adeno carcinoma,

Adeno-squamous carcinoma or AIS we want to examine prospectively:

1. Examine if negative HR-HPV after conization to the HR-HPV the women had before conization has a high prognostic value for no residual tumor in the final pathology.
2. To examine if conization in women with cervical tumor up to Stage I B 2 (FIGO 2018) is corelated with better prognosis.

DETAILED DESCRIPTION:
The treatment of invasive cervical cancer is tailored according to the FIGO recommendations. The standard treatment for women with early-stage, (IA2-IB1) cervical cancer is simple or Radical Hysterectomy (RH) and in women with Adenocarcinoma in Situ hysterectomy is recommended when they finish their fertility program .A Few studies describe that conization before Radical Hysterectomy in women with cervical cancer stage I B 1 ( tumour up to 4 cm according to FIGO 2009 ) , are in correlation with better prognosis , Bizzari describe women that had conization before RH had better 5 year survival. Uppal report that those women have less recurrence, OR of 0.4 compared with women without conization. Chacon summarize SUCCOR study, a multi center study that collected data about 374 women with cervical cancer Stage I B 1 according to FIGO 2009 -tumour up to 4 cm .187 women had conization before RH and 187 had RH without conization. Women that had conization had 65% less recurrence 'and 75% les mortality.

Several studies have explored the possibility of a less aggressive approach for cervical cancer patients with low-risk early-stage disease who wish to preserve fertility. The parameters that were investigated were: the depth of invasion, tumour diameter, lymph node status positive margins in conization, positive Endo Cervical Curettage (ECC) and lymph-vascular space invasion. Those parameters have a low sensitivity and between 50-65% of women who had RH had no residual tumour in the final pathology.

Schmeler describe that woman who had conization before RH in 97.5% had no residual tumour.

A study of 92 women with cervical cancer and Adeno Carcinoma In situ (AIS) that short time after conization were negative to High-Risk HPV (HR-HPV) they had before the conization in 95% there was no residual tumour in the final pathology, or during the follow up.

To our knowledge there is no prospective study that examined the the prognostic value of Conization and negative HR- HPV typing after Conization prior to surgical intervention in Early-Stage Cervical Cancer and Adenocarcinoma in Situ.

Aim:

In women with cervical cancer -Squamous cell carcinoma, Adeno carcinoma,

Adeno-squamous carcinoma or AIS we want to examine prospectively:

1. Examine if negative HR-HPV after conization to the HR-HPV the women had before conization has a high prognostic value for no residual tumour in the final pathology.
2. To examine if conization in women with cervical tumour up to Stage I B 2 (FIGO 2018) is corelated with better prognosis.

ELIGIBILITY:
Inclusion Criteria:

Age Range: 18-85 years old Cervical cancer stage I B 2(Tumor up to 4 cm FIGO 2018) AIS HPV types before and after conization

Exclusion Criteria:

Pregnant women under 18 years old. Women who refused to continue to be in study. Women that data about HPV types , final pathology or complication are missing.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with cervical cancer -Squamous cell carcinoma, Adeno carcinoma, Adeno-squamous carcinoma or AIS
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Final Pathology | 1 year
  Residual disease in final pathology

SECONDARY OUTCOMES:
Disease recurrence | 5 year
  number of months until Disease recurrence
Mortality | 5 year
  mortality rate during the study between the groups
complications | 5 year
  major complications

CONTACTS AND LOCATIONS:
Overall Officials: Yoav Siegler, MD, Principal Investigator — Rambam Health Care Center
Locations (1):
- Rambam Health Care Center, Haifa, Israel

REFERENCES:
- [Background] de Sanjose S, Quint WG, Alemany L, Geraets DT, Klaustermeier JE, Lloveras B, Tous S, Felix A, Bravo LE, Shin HR, Vallejos CS, de Ruiz PA, Lima MA, Guimera N, Clavero O, Alejo M, Llombart-Bosch A, Cheng-Yang C, Tatti SA, Kasamatsu E, Iljazovic E, Odida M, Prado R, Seoud M, Grce M, Usubutun A, Jain A, Suarez GA, Lombardi LE, Banjo A, Menendez C, Domingo EJ, Velasco J, Nessa A, Chichareon SC, Qiao YL, Lerma E, Garland SM, Sasagawa T, Ferrera A, Hammouda D, Mariani L, Pelayo A, Steiner I, Oliva E, Meijer CJ, Al-Jassar WF, Cruz E, Wright TC, Puras A, Llave CL, Tzardi M, Agorastos T, Garcia-Barriola V, Clavel C, Ordi J, Andujar M, Castellsague X, Sanchez GI, Nowakowski AM, Bornstein J, Munoz N, Bosch FX; Retrospective International Survey and HPV Time Trends Study Group. Human papillomavirus genotype attribution in invasive cervical cancer: a retrospective cross-sectional worldwide study. Lancet Oncol. 2010 Nov;11(11):1048-56. doi: 10.1016/S1470-2045(10)70230-8. Epub 2010 Oct 15. PMID 20952254
- [Background] Siegler E, Reichman Y, Kugelman N, Mackuli L, Lavie O, Ostrovsky L, Shaked-Mishan P, Segev Y. Low-Risk Human Papillomavirus Types in Cervical Intraepithelial Neoplasia 2-3 and in Invasive Cervical Cancer Patients. J Low Genit Tract Dis. 2019 Oct;23(4):248-252. doi: 10.1097/LGT.0000000000000486. PMID 31592971
- [Background] Cuschieri K, Bhatia R, Cruickshank M, Hillemanns P, Arbyn M. HPV testing in the context of post-treatment follow up (test of cure). J Clin Virol. 2016 Mar;76 Suppl 1:S56-S61. doi: 10.1016/j.jcv.2015.10.008. Epub 2015 Oct 22. PMID 26525202
- [Background] Bizzarri N, Pedone Anchora L, Kucukmetin A, Ratnavelu N, Korompelis P, Carbone V, Fedele C, Bruno M, Vizzielli G, Gallotta V, De Vincenzo R, Chiantera V, Fagotti A, Fanfani F, Ferrandina G, Scambia G. Protective Role of Conization Before Radical Hysterectomy in Early-Stage Cervical Cancer: A Propensity-Score Matching Study. Ann Surg Oncol. 2021 Jul;28(7):3585-3594. doi: 10.1245/s10434-021-09695-4. Epub 2021 Feb 23. PMID 33620615
- [Background] Uppal S, Gehrig PA, Peng K, Bixel KL, Matsuo K, Vetter MH, Davidson BA, Cisa MP, Lees BF, Brunette LL, Tucker K, Stuart Staley A, Gotlieb WH, Holloway RW, Essel KG, Holman LL, Goldfeld E, Olawaiye A, Rose SL. Recurrence Rates in Patients With Cervical Cancer Treated With Abdominal Versus Minimally Invasive Radical Hysterectomy: A Multi-Institutional Retrospective Review Study. J Clin Oncol. 2020 Apr 1;38(10):1030-1040. doi: 10.1200/JCO.19.03012. Epub 2020 Feb 7. PMID 32031867
- [Background] Chacon E, Manzour N, Zanagnolo V, Querleu D, Nunez-Cordoba JM, Martin-Calvo N, Capilna ME, Fagotti A, Kucukmetin A, Mom C, Chakalova G, Shamistan A, Gil Moreno A, Malzoni M, Narducci F, Arencibia O, Raspagliesi F, Toptas T, Cibula D, Kaidarova D, Meydanli MM, Tavares M, Golub D, Perrone AM, Poka R, Tsolakidis D, Vujic G, Jedryka MA, Zusterzeel PLM, Beltman JJ, Goffin F, Haidopoulos D, Haller H, Jach R, Yezhova I, Berlev I, Bernardino M, Bharathan R, Lanner M, Maenpaa MM, Sukhin V, Feron JG, Fruscio R, Kukk K, Ponce J, Minguez JA, Vazquez-Vicente D, Castellanos T, Boria F, Alcazar JL, Chiva L; SUCCOR study group; SUCCOR study Group. SUCCOR cone study: conization before radical hysterectomy. Int J Gynecol Cancer. 2022 Feb;32(2):117-124. doi: 10.1136/ijgc-2021-002544. Epub 2022 Jan 17. PMID 35039455
- [Background] Plante M, Renaud MC, Francois H, Roy M. Vaginal radical trachelectomy: an oncologically safe fertility-preserving surgery. An updated series of 72 cases and review of the literature. Gynecol Oncol. 2004 Sep;94(3):614-23. doi: 10.1016/j.ygyno.2004.05.032. PMID 15350349
- [Background] Suri A, Frumovitz M, Milam MR, dos Reis R, Ramirez PT. Preoperative pathologic findings associated with residual disease at radical hysterectomy in women with stage IA2 cervical cancer. Gynecol Oncol. 2009 Jan;112(1):110-3. doi: 10.1016/j.ygyno.2008.09.011. Epub 2008 Oct 25. PMID 18952270
- [Background] Li X, Xia L, Chen X, Fu Y, Wu X. Simple conization and pelvic lymphadenectomy in early-stage cervical cancer: A retrospective analysis and review of the literature. Gynecol Oncol. 2020 Aug;158(2):231-235. doi: 10.1016/j.ygyno.2020.05.035. Epub 2020 Jun 6. PMID 32518013
- [Background] Costa S, Negri G, Sideri M, Santini D, Martinelli G, Venturoli S, Pelusi C, Syrjanen S, Syrjanen K, Pelusi G. Human papillomavirus (HPV) test and PAP smear as predictors of outcome in conservatively treated adenocarcinoma in situ (AIS) of the uterine cervix. Gynecol Oncol. 2007 Jul;106(1):170-6. doi: 10.1016/j.ygyno.2007.03.016. Epub 2007 May 4. PMID 17481701
- [Background] Costa S, Sideri M, Negri G, Venturoli S, Santini D, Casadio C, Sandri MT, Bucchi L. The predictive value of human papillomavirus testing for the outcome of patients conservatively treated for stage IA squamous cell cervical carcinoma. J Clin Virol. 2015 Sep;70:53-57. doi: 10.1016/j.jcv.2015.07.007. Epub 2015 Jul 8. PMID 26305820
- [Background] Siegler E, Goldberg Y, Siegler Y, Shaked-Mishan P, Mazareb S, Kugelman N, Mackuli L, Sabo E, Lavie O, Segev Y. The Association Between Clearance of Human Papillomavirus After Conization for Cervical Cancer and Absence of Cancer. J Low Genit Tract Dis. 2021 Oct 1;25(4):276-280. doi: 10.1097/LGT.0000000000000622. PMID 34369434